CLINICAL TRIAL: NCT03874468
Title: Prevalence of Coronal Femoral Bowing in the Egyptian Arthritic Knee
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kerolos Naiem Shehata Rofael (Other)
Responsible Party: Sponsor-Investigator, Kerolos Naiem Shehata Rofael, Principle investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: coronal femoral Bowing
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Arthritis Knee
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: X-ray — standing anteroposterior radiographs of the full-length lower limb with patients in the standing position. ( HKA Long Film Radiographs ).

SUMMARY:
To Detect the Prevalence Of Coronal Femoral Bowing in Egyptian arthritic knee. The restoration of normal coronal alignment of the lower extremity is very important to surgeons who perform reconstructive surgery of the knee, such as total knee arthroplasty (TKA). The importance of achieving normal coronal alignment of the lower extremity after TKA is widely recognized . TKAs with coronal malalignment tend to fail earlier than those with neutral alignment. 8 Coronal alignment is considered key to the function and longevity of a TKA. However, most studies do not consider femoral and tibial anatomical features such as coronal femoral bowing and the effects of these features and subsequent alignment on function after TKA are unclear investigators therefore determined the prevalence of coronal femoral bowing, femoral condylar orientation (mLDFA ) , and tibia plateau inclination (mMPTA ) in osteoarthritic Egyptian population

DETAILED DESCRIPTION:
Radiological methods :

1) standing anteroposterior radiographs of the full-length lower limb with patients in the standing position. ( HKA Long Film Radiographs ).

Measurements :

1. mechanical hip-knee-ankle axis (HKA) angle: the angle formed by the mechanical axes of the femur and tibia
2. anatomical hip-knee-ankle axis (HKA) angle: the angle formed by the anatomical axes of the femur and tibia
3. For condylar orientation : the mechanical lateral distal femoral angle (mLDFA) was defined as an angle formed by the mechanical axis of the femur and the line connecting the distal ends of the medial and lateral femoral condyles of the femur.
4. For tibia plateau inclination : the mechanical lateral proximal tibial angle (mLPTA) was defined as an angle formed by the mechanical axis of the tibia and the articular surface of the proximal tibia .
5. Coronal femoral bowing Using the method of Yau et al. : the femoral diaphysis was divided into four equal parts, . Because Yau et al. didn't exactly describe the femoral diaphysis, we had defined the femoral diaphysis from the lower border of the lesser trochanter to upper border of the distal femoral segment which is defined by a square whose sides have the same length as the widest part of the femoral condyle so called rule of square (from the lowest level of the lesser trochanter to 5 cm above the lowest level of the lateral femoral condyle), and the midpoint of the endosteal intramedullary canal was depicted in each quarter. The angulation between midlines drawn in the proximal and distal quarters of the femoral diaphysis will be measured

ELIGIBILITY:
Inclusion Criteria:

-Any advanced Osteoarthritic patient schedual for TKA

Exclusion Criteria:

* History of femoral or tibial fracture or osteotomy around the knee .
* Presence of a congenital anomaly in the femur or tibia .
* History of prior knee or hip arthroplasty .
* Diagnosis other than primary osteoarthritis (RA-inflmmatory arthritis..etc) .
* Position in radiographs preventing complete evaluation of radiographic variables .

Ages: 20 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: any Egyptian patient who suffer from advanced osteoarthritis schedual for TKR at any age ,any sex
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
To asses the Prevalence Of Coronal Femoral Bowing in Egyptian arthritic knee | Baseline
  Coronal Femoral Bowing in Egyptian arthritic knee may be prevalent and its effect on TKR will be measured and reported

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kobayashi H, Akamatsu Y, Kumagai K, Kusayama Y, Aratake M, Saito T. Influence of coronal bowing on the lower alignment and the positioning of component in navigation and conventional total knee arthroplasty. Orthop Traumatol Surg Res. 2017 Apr;103(2):251-256. doi: 10.1016/j.otsr.2016.11.017. Epub 2017 Jan 11. PMID 28087396
- [Background] Nakano N, Matsumoto T, Hashimura M, Takayama K, Ishida K, Araki D, Matsushita T, Kuroda R, Kurosaka M. Coronal lower limb alignment in normal knees--A radiographic analysis of 797 normal knee subjects. Knee. 2016 Mar;23(2):209-13. doi: 10.1016/j.knee.2015.12.004. Epub 2016 Jan 7. PMID 26775257